CLINICAL TRIAL: NCT07246473
Title: Study on the Safety and Efficacy of Non-Invasive Transcranial Doppler Ultrasound in Promoting Hematoma Clearance for Intracerebral Hemorrhage
Brief Title: Non-invasive Ultrasound and Hematoma Clearance After Intracerebral Hemorrhage
Acronym: NOTICE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruijun Ji, Chief Physician/Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFH-brain2024-2-2051
Record Dates: First submitted 2025-09-23; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Intervention Group (Experimental): On the basis of best medical management, 2 MHz non-invasive ultrasonic scalpel was used for intervention within 48-72 hours after the occurrence of intracerebral hemorrhage, 20min/ day, and continued for 7 days.
  Interventions: Device: non-invasive ultrasonic scalpel
- Sham Comparator (Sham Comparator): On the basis of best medical management, a sham non-invasive ultrasonic scalpel (simulating real treatment with zero energy output) was applied within 48-72 hours after the occurrence of intracerebral hemorrhage, 20 min/day for 7 consecutive days
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: non-invasive ultrasonic scalpel — On the basis of best medical management, 2 MHz non-invasive ultrasonic scalpel was used for intervention within 48-72 hours after the occurrence of intracerebral hemorrhage, 20min/ day, and continued for 7 days.
  Arms: Ultrasound Intervention Group
Device: Sham Comparator — On the basis of best medical management, a sham non-invasive ultrasonic scalpel (simulating real treatment with zero energy output) was applied within 48-72 hours after the occurrence of intracerebral hemorrhage, 20 min/day for 7 consecutive days
  Arms: Sham Comparator

SUMMARY:
Intracerebral hemorrhage (ICH) is one of the stroke subtypes with the highest global rates of disability and mortality, accounting for 15%-20% of all strokes. Currently, there is a lack of evidence-based interventions for ICH, with treatment primarily relying on supportive care. There is an urgent clinical need to explore new strategies and technologies. The investigators hypothesize that for ICH patients, best medical treatment combined with a non-invasive ultrasonic scalpel (ultrasound Doppler flow analyzer) may be superior to best medical treatment alone. The primary objective of this study is to determine the safety and efficacy of the non-invasive ultrasonic scalpel in promoting hematoma clearance in ICH patients.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, controlled trial investigating the use of a 2MHz non-invasive ultrasonic scalpel (ultrasound Doppler flow analyzer, registered as Medical System for Ultrasound Diagnosis) in patients with acute ICH. Eligible participants (n=86 will be randomized 1:1 to either the intervention group (ultrasound + standard medical treatment) or the control group (sham ultrasound + standard treatment). The ultrasound intervention involves daily 20-minute sessions for 7 consecutive days. Primary outcomes include hematoma clearance rates and neurological function improvement, assessed via imaging and clinical scales at multiple time points (baseline, 24±12 hours, 72±12 hours, 7±1days/discharge, 3 months). Safety will be monitored through adverse event tracking, vital signs, and neurological examinations. Ethical approval has been obtained, and all participants will provide informed consent. The trial is conducted at Beijing Tiantan Hospital, with results expected to advance non-invasive ICH treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years;
* Spontaneous intracerebral hemorrhage (ICH);
* Supratentorial ICH;
* Hematoma volume <30 mL (calculated using the ABC/2 method);
* Glasgow Coma Scale (GCS) score >9 at randomization;
* Time from onset to randomization: 48-72 hours;
* Patient and/or legal representative provides informed consent.

Exclusion Criteria:

* Intracerebral hemorrhage attributed to other causes (e.g., cerebral aneurysm, cerebrovascular malformation, brain tumor, cerebral venous sinus thrombosis, hemorrhagic transformation of ischemic stroke, head trauma, anticoagulation therapy, hematologic disorders).
* Hemorrhage located in the infratentorial region.
* Hemorrhage confined primarily to the ventricular system.
* Clinical signs or symptoms suggestive of brain herniation (e.g., progressive decline in level of consciousness, diminished or absent pupillary light reflexes, bilateral pyramidal signs).
* Severe cardiac dysfunction (NYHA Class III or IV).
* High-risk chronic arrhythmias (e.g., sick sinus syndrome, second- or third-degree atrioventricular block, bradycardia-related syncope without pacemaker implantation).
* Severe hepatic impairment defined as ALT >2x ULN or AST >2x ULN (ULN = Upper Limit of Normal).
* Severe renal impairment defined as serum creatinine >1.5x ULN.
* History of severe asthma or chronic obstructive pulmonary disease (COPD).
* History of coagulopathy or systemic bleeding disorder.
* Leukopenia (<2 × 10⁹/L) or thrombocytopenia (<100 × 10⁹/L).
* Patients scheduled for surgical intervention (including, but not limited to, hematoma evacuation [minimally invasive or conventional], decompressive craniectomy, hematoma aspiration, or external ventricular drainage) prior to the first dose of study treatment.
* Pre-stroke modified Rankin Scale (mRS) score >2.
* Presence of other severe disease resulting in a life expectancy of less than 1 year.
* Inability to understand the study procedures and/or complete follow-up due to psychiatric illness, cognitive impairment, or emotional disorders.
* Women who are pregnant or lactating.
* Participation in another clinical trial within the past 3 months or current participation in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematoma clearance rate on CT at Day 7±1day after randomization/discharge； | Day 7±1day after randomization/discharge
  Hematoma clearance rate is defined as the percentage reduction in intracerebral hematoma volume from baseline to the follow-up CT scan. It is calculated using the formula: [(Baseline volume - Follow-up volume) / Baseline volume] x 100%.

SECONDARY OUTCOMES:
Hematoma expansion on CT at 24±12 hours after randomization | 24±12 hours after randomization
  A relative increase in hematoma volume ≥ 33%, calculated as: (Follow-up volume - Baseline volume) / Baseline volume ≥ 33%; OR An absolute increase in hematoma volume ≥ 12.5 mL, calculated as: Follow-up volume - Baseline volume ≥ 12.5 mL；
Neurological improvement at 24±12 hours after randomization (NIHSS(baseline)- NIHSS(24±12 hours)) | 24±12 hours after randomization
  Neurological status as assessed by the National Institutes of Health Stroke Scale (NIHSS) score； The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. The scale ranges from 0 to 42, where a higher score indicates more severe neurological deficit.
Absolute hematoma volume (mL) on CT at 72±12 hours after randomization | 72±12 hours after randomization
Neurological improvement at 72±12 hours after randomization(NIHSS(baseline)- NIHSS(72±12 hours)) | 72±12 hours after randomization
  Neurological status as assessed by the National Institutes of Health Stroke Scale (NIHSS) score； The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. The scale ranges from 0 to 42, where a higher score indicates more severe neurological deficit.
Absolute hematoma volume (mL) on CT at Day 7±1day after randomization/discharge | Day 7±1 day after randomization or discharge
Absolute perihematomal edema (PHE) volume (mL) on CT at Day 7±1day after randomization/discharge | Day 7±1 day after randomization or discharge
Neurological improvement at Day 7±1day after randomization/discharge(NIHSS(baseline)- NIHSS( Day 7±1day)) | Day7±1day after randomization or discharge
  Neurological status as assessed by the National Institutes of Health Stroke Scale (NIHSS) score； The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. The scale ranges from 0 to 42, where a higher score indicates more severe neurological deficit.
Modified Rankin Scale (mRS) score at 90±7 days after onset | 90±7 days after onset
  The modified Rankin Scale (mRS) is a standardized measure of global functional outcome and degree of disability or dependence after a stroke or other neurological disorder. It is a 7-point scale ranging from 0 to 6, with specific criteria for each grade:
  0 - No symptoms at all.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead. A lower score indicates a better functional outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ruijun Ji, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No